CLINICAL TRIAL: NCT02772705
Title: Comparison of Standardized Update Value Using Single-photo Emission Computed Tomography and Computed Tomography Between Grave's Disease (Hyperthyroidism) Patients and Normal Humans
Brief Title: Comparison of SUV Using SPECT/CT Between Grave's Disease Patients and Normal Humans
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Guangzhou Panyu Central Hospital (Other); Hebei General Hospital (Other); Air Force Military Medical University, China (Other); Zhejiang Cancer Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Li Yuhao, Technologist, a graduated student of Department of Nuclear Medicine, West China Hospital
Other Study IDs: 2016-92
Record Dates: First submitted 2016-05-09; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Hyperthyroidism; Tomography; Emission-Computed; Single-Photon
Keywords: Standardized Uptake Value; Diagnosis
MeSH Terms: conditions — Hyperthyroidism; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hyperthyroidism: Those with Grave's Disease(GD,Hyperthyroidism),with lower TSH, and higher FT3, FT4.
- Health Humans: Those humans who are healthy, without GD, without any treatment, with normal TSH, FT3, FT4.

SUMMARY:
The purpose of this study is to find out the capacity of standardized uptake value (SUV) using single-photo emission computed tomography and computed tomography (SPECT/CT) in diagnosing Grave's Disease (hyperthyroidism).

DETAILED DESCRIPTION:
Traditionally it is considered that only positron emission tomography(PET) has the ability to obtain standardized uptake value（SUV）while single-photo emission computed tomography(SPECT) does not have. Recently with the developing of technology, the ability of SPECT has been extended.

On the other hand, thyroid imaging by SPECT can only play an auxiliary role in hyperthyroidism diagnosis mainly since it is regarded as nonquantitative. So the investigators design this study to search the capacity and accuracy of SUV provided by SPECT and CT(CT is used for reconstruction algorithm) in diagnosing GD.

This is a multiple-center study containing nine groups in China that use GE Discovery NM/CT, an advanced equipment. Thus, the data can be more accurate and more available.

And this is a perspective clinical trial, taking about eight months. The investigators plan to evaluate at least 50 Grave's Disease(GD) patients and 50 normal humans as contrast in all.

Every GD patient must have been diagnosed and the results of thyroid function tests(such as TSH,FT3,FT4） must be available. If necessary, the patient's rate of iodine uptake should also be known before he/she being included in this study. As for normal people, the results of thyroid function tests should be within the range of normal value.

The data of each participant will be gathered and stored. And the data processing will be done with the help of GE staff, using the software Q.Metrix to get the value of SUVmean, SUVmax. Finally T test will be used in comparison of the differences.

ELIGIBILITY:
For Group of GD Patients:

Inclusion Criteria:

* certainly diagnosed with GD
* no treatment
* sign a informed consent

Exclusion Criteria:

* Inflammatory Hyperthyroidism
* Secondary Hyperthyroidism (since of medicine, thyrotrophs neoplasms and etc)
* Can not finish the check of SPECT/CT
* Refuse to sign a informed consent

For Group of Normal Humans:

Inclusion Criteria:

* without GD
* Adult
* sign a reformed consent

Exclusion Criteria:

* Without normal values of TSH, FT3, FT4
* Can not finish the check of SPECT/CT
* Failed to sign a reformed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As for GD patients, the study samples will be chosen from the patients in every medical center which participates in this study. And they will be chosen before their treatment.
  For the normal humans, they are healthy volunteers without thyroid disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-08 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
The thyroid imaging of GD patients and normal humans by SPECT/CT | a single point in time, at subject enrollment
  For GD patients and normal healthy volunteers, we will get the data of thyroid fusion imaging by giving them a SPECT/CT check at subject enrollment.
The SUV values of GD patients and normal humans provided by Q.Metrix | a single point in time, at subject enrollment
  The data of thyroid fusion imaging will be processed by the software, Q.Metrix, which can get the accurate SUV by compensating for photon absorption within the body, removing scattered radiation and etc.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Li, Master, Study Chair — West China Hospital of Sichuan University, Department of Nuclear Medicine; Xiaohong Ou, Ph.D, Study Director — West China Hospital of Sichuan University, Department of Nuclear Medicine; Yahao Li, Bachelor, Principal Investigator — West China Hospital of Sichuan University, Department of Nuclear Medicine
Locations (9):
- China (9):
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - Guangzhou Panyu Central Hospital, Guangzhou, Guangdong
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The People's Hospital of Inner Mongolia Autonomous Region, Hohhot, Inner Mongolia
  - Fourth Military Medical Universit, Xi’an, Shanxi
  - West China Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
The data of the subjects will be shared including gender, age, values of SUV, TSH, FT3, FT4 and other relative records.
  The information will not be shared until the study is completed and the article is published.
  Anyone who wants to get the data should send an e-mail to Li, with reasons for needing these data.
  E-mail address: 617381606@qq.com

REFERENCES:
- [Background] Bailey DL, Willowson KP. An evidence-based review of quantitative SPECT imaging and potential clinical applications. J Nucl Med. 2013 Jan;54(1):83-9. doi: 10.2967/jnumed.112.111476. PMID 23283563